## Joint Position Sense in Individuals with Anterior Knee Pain

<u>Informed consent form</u> <u>Document date: 19/6/2019</u>

Carlyn Rhode (BSc Physiotherapy, MPhysiotherapy), Postgraduate student at
Stellenbosch University; Quinette Louw (BSc Physiotherapy, MPhysiotherapy, PhD
Physiotherapy), Professor of Physiotherapy at Stellenbosch University; Dominique
Leibbrandt (BSc Physiotherapy, MPhysiotherapy, PhD Physiotherapy), Post-doctoral
researcher at Stellenbosch University; Leoné Williams (BSc Physiotherapy,
MPhysiotherapy), Lecturer at Stellenbosch University

Faculty of Medicine and Health Sciences – University of Stellenbosch,

Physiotherapy Division/FNB-3D Movement Analysis Laboratory,

PO Box 19063 / Francie van Zijl Drive, Tygerberg 7505, South Africa.

Participant Information Leaflet and Consent Form
TITLE OF THE RESEARCH PROJECT: Proprioception changes in individuals with
Anterior knee pain.

PRINCIPAL INVESTIGATOR: Carlyn Rhode

ADDRESS: Faculty of Medicine & Health Sciences, Division of Physiotherapy,

Stellenbosch University, 4th floor, Teaching Building, Tygerberg, 7505

**CONTACT NUMBER: 021 938 9667** 

You are being invited to partake in a research project. Please take some time to read the information presented here, which will explain the details of this project. Please ask the study staff or doctor any questions about any part of this project that you do not fully understand. It is very important that you are fully satisfied that you clearly understand what this research entails and how you could be involved. Also, your participation is entirely voluntary and you are free to decline to participate. If you say no, this will not affect you negatively in any way whatsoever. You are also free to withdraw from the study at any point, even if you do agree to take part.

This study has been approved by the Health Research Ethics Committee of Stellenbosch
University and will be conducted according to the ethical guidelines and principles of the
international Declaration of Helsinki, South African Guidelines for Good Clinical Practice and the
Medical Research Council (MRC) Ethical Guidelines for Research.

#### What is this research study all about?

Adolescents and young adults often experience pain in front of the knee, referred to as a condition called anterior knee pain. The cause and factors contributing to pain in front of the knee are still unknown.

The purpose of this research project is to determine whether people with pain in front of the knee have difficulty in sensing the precise position of their knee joint during movement (this

sense of position is called proprioception). This study will take place at the FNB-3D movement analysis clinic, Stellenbosch University, Tygerberg Medical School Campus. This project will include 30 individuals, aged between 14 and 40 years who experience anterior knee pain. Participants will be assessed for anterior knee pain by the senior physiotherapist at the FNB-3D movement analysis clinic. Reflective markers will be placed on bony landmarks of the lower limb to allow the researcher to evaluate the affected knees sense of position. Each participant will perform 3 active knee tests movements in 3 different test positions; Extending the knee in sitting, bending the knee in prone and single leg squat in standing in a full weight- bearing position. The duration of testing is 90 minutes. We will also measure your height, weight, leg length and other body dimensions.

All these procedures are non-invasive. Participants will be carefully instructed and guided through each test position and a practice trial just to familiarize them with the test movements. Participants will be blindfolded at the commencement of testing to prevent any visual guiding during testing. We will also measure the intensity of your knee pain and functional problems using questionnaires.

#### Why have you been invited to participate?

You have been invited to participate in this the study because you experience anterior knee pain and responded to our invitations or advertisements.

What will your responsibilities be?

You will be required pay a once-off visit to the FNB-3D movement analysis clinic for knee testing.

#### Will you benefit from taking part in this research?

You will contribute to updating the evidence on anterior knee pain. The knowledge gained may help to improve future rehabilitation of persons with anterior knee pain.

Are there in risks involved in your taking part in this research?

There is a small risk that you may develop a skin reaction due to the electrodes. This skin reaction will settle within a day or two and will usually not require treatment.

If you do not agree to take part, what alternatives do you have?

You can receive treatment, at your own cost, at the FNB-3D movement analysis clinic or, at any other therapist of your choice.

#### Who will have access to your medical records?

All information obtained from you will be treated as strictly confidential. Only the researchers involved in the study will have access to the data collected.

We will publish the findings of the study in a scientific journal and will also present it at scientific meetings/conferences; anonymity of your identity will be maintained.

# What will happen in the unlikely event of some form injury occurring as a direct result of your taking part in this research study?

The university's indemnity insurance will cover the cost of any unfortunate incidents incurred during the testing procedures.

Will you be paid to take part in this study and are there any costs involved?

No but you will be reimbursed for your time and travel costs with an amount of R200. There are no cost involved for taking part in the study.

#### Is there anything else that you should know or do?

Ø You can contact Prof Q. Louw at tel 021 9389667 if you have any further queries or encounter any problems.

Ø You can contact the Health Research Ethics Committee at 021-938 9207 if you have any concerns or complaints that have not been adequately addressed by your study physiotherapist.

 $\emptyset$  You will receive a copy of this information and consent form for your own records.

### **Declaration by participant**

By signing below, I ...... agree to take part in a research study entitled (Is proprioception affected in individuals with anterior knee pain?)

I declare that:

- I have read or had read to me this information and consent form and it is written in a language with which I am fluent and comfortable.
- I have had a chance to ask questions and all my questions have been adequately answered.
- I understand that taking part in this study is voluntary and I have not been pressurized to take part.
- I may choose to leave the study at any time and will not be penalized or prejudiced in any way.
- I may be asked to leave the study before it has finished, if the study doctor or researcher feels it is in my best interests, or if I do not follow the study plan, as agreed to.

| Signed at (place) | on (date) | 2017 |
|------------------------------------|---------------|------|
| Signature of participant Signature | of witness | |
| Declaration by investigator | | |
| I (name) | declare that: | |

- I explained the information in this document to .....
- I encouraged him/her to ask questions and took adequate time to answer them.
- I am satisfied that he/she adequately understands all aspects of the research, as discussed above
- I did/did not use an interpreter. (If an interpreter is used then the interpreter must sign the declaration below.

| Signed at (place) | on | (date) 2017. |
|-------------------|----|--------------|

Signature of investigator Signature of witness